CLINICAL TRIAL: NCT06658132
Title: An Exploratory Study of a General Anesthesia Regimen for Deep Brain Electrical Stimulation in Patients With Parkinson's Disease
Brief Title: A General Anesthesia Regimen for DBS Surgery in Patients With PD
Acronym: GADBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Jie Tian, Principal Investigator, RenJi Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Anesthesia Methods for DBS
Record Dates: First submitted 2024-10-23; First posted 2024-10-26 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Parkinson's Disease (PD)
Keywords: deep brain electrical stimulation; a general anesthesia regimen; esketamine; remifentanil; Parkinson's disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- remifentanil combined with esketamine (Experimental): a novel anesthesia regimen of remifentanil combined with esketamine for the physiological testing phase of DBS surgery.
  Interventions: Drug: 0.5~1ug/kg/min remifentanil combined with 0.2~0.5mg/kg/h esketamine for the physiological testing phase of DBS surgery.

INTERVENTIONS:
Drug: 0.5~1ug/kg/min remifentanil combined with 0.2~0.5mg/kg/h esketamine for the physiological testing phase of DBS surgery. — Throughout the first and third stages of surgery, all patients receive a traditional induction of anesthesia. Fifteen minutes before the second stage of surgery (MER and clinical assessment), when the burr hole is ready, the propofol and sevoflurane infusion is discontinued, and patients receive 0.5~1ug/kg/min remifentanil combined with 0.2~0.5mg/kg/h esketamine. On completion of the second stage of surgery, the interventional drug is discontinued and propofol combined with sevoflurane is resumed until the end of the third stage.

SUMMARY:
Patients who meet the enrollment criteria and voluntarily join this study will be admitted to the operating room on the day of surgery, and will receive endotracheal intubation under general anesthesia. Induction will be conducted with sufentanil 0.2~0.3ug/kg, rocuronium bromide 0.6mg/kg and propofol 1~2 mg/kg. After successful intubation, mechanical ventilation will be provided with a fresh air flow of 2.0 L/min, a tidal volume of 6~8ml/kg and a respiratory rate of 10~12 times/min to control the end-tidal carbon dioxide between 35~45mmHg. Following that, 20 ml of 0.5% ropivacaine will be applied for bilateral scalp nerve block. The surgeon will then install the stereotactic head frame and take the patients out for CT examination. After returning to the operating room after CT examination, the surgeons will install driving electrodes. During this period, GA will be maintained with sevoflurane, propofol, remifentanil and rocuronium bromide. The depth of anesthesia is monitored using BIS, with a target of 40-65.

During electrode implantation stage: sevoflurane, propofol and rocuronium bromide will be stopped, and esketamine 0.2~0.5mg/kg/h combined with remifentanil 0.5~1ug/kg/min will be used to maintain anesthesia with a target BIS value of 60-70. Patients' blood pressure and heart rate will be controlled to change within less than 30% of the basal value with necessary medication.

If the patient moves during the electrode implantation stage, the rescue plan is to quickly inhale sevoflurane to 0.3 mac, and the number of rescues will be recorded. The vital signs of the patient, MER signal strength, STN discharge frequency, length of STN localization nucleus, and whether the STN boundary is successfully located will be recorded.

During the implantation stage of the pulser, the GA regimen will return to before electrode implantation stage. In other words, sevoflurane + remifentanil + propofol + rocuronium bromide will be used to maintain the depth of anesthesia till the end of the operation.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral STN-DBS surgery is planned for primary PD (meeting the International Movement Disorder Society (MDS) diagnostic criteria for PD);
* ASA Classes I-III;
* Age 50-75 years;
* Informed consent from patients or their families

Exclusion Criteria:

* BMI≥28.0kg/m2；
* comorbid other conditions causing parkinson-like motor symptoms;
* Previous history of severe head trauma, deformity, or craniocerebral surgery;
* Previous history of psychiatric and neurological diseases, such as history of overt stroke (ischemic lesion near STN), depression, severe central nervous system depression, basal gangliopathy, schizophrenia, epilepsy, Alzheimer's disease, myasthenia gravis, etc.;
* Preoperative MoCA scale showed that the patient had dementia;
* Severe heart, liver, lung, kidney, and immune system diseases;
* Allergy or contraindication to the trial drug

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-10-29 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Proportion of MER signal recordings with high NRMS. | During surgery
  Mean NRMS greater than 2.0 after MER recording after STN entry.

SECONDARY OUTCOMES:
MER signal strength | During surgery
Beta band (13-30Hz) oscillations calculated by spectrum analysis during MER recording. | During surgery
Length of STN | During surgery
Proportion of successfully defining STN borders | During surgery
occurrence of cognitive impairment at 7 days postoperatively | at 7 days postoperatively
  MoCA scale score decreased by 2 points compared with preoperatively
occurrence of depression at 7 days postoperatively | at 7 days postoperatively
  HAMD scale score> 20 points
Patient satisfaction at 24 hours after surgery | at 24 hours after surgery
  Analyzed by patient satisfaction assessment scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China